CLINICAL TRIAL: NCT07242755
Title: The Effect of Crossword Puzzle Activity on Nursing Students' Knowledge Level Regarding Safe Medication Practices: A Randomized Controlled Trial
Brief Title: Crossword Puzzle Activity on Students' Knowledge Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gulden Basit, Dr, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GIU-2025-26
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Knowledge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- crossword puzzle (Experimental): In addition to theoretical topics, the intervention group will participate in a puzzle activity related to the topic covered in the course for 7 weeks.
  Interventions: Other: active learning method (crossword puzzle)
- control (No Intervention): The control group will receive standard theoretical training.

INTERVENTIONS:
Other: active learning method (crossword puzzle) — Students in the intervention group will participate in a crossword puzzle activity, which is one of the active learning methods.
  Arms: crossword puzzle

SUMMARY:
The purpose of this study was to evaluate the effect of a crossword puzzle activity designed for nursing students on their knowledge levels regarding safe medication practices. Students will be divided into two groups: the intervention group will complete a course-related crossword puzzle activity, and the control group will receive standard theoretical instruction.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of a crossword puzzle activity designed for nursing students on their knowledge levels regarding safe medication practices. Students will be divided into two groups: the intervention group will complete a course-related crossword puzzle activity for seven weeks, and the control group will receive standard theoretical instruction.Students will be randomly assigned to groups. A knowledge test on safe medication practices will be administered before the intervention and at the end of the 7-week period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being in the final year of nursing
* Taking the safe medication practices course for the first time

Exclusion Criteria:

* Being a foreign national and having problems reading and understanding Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Nursing Students' Knowledge Level Regarding Safe Medication Practices | at the end of the seven weeks
  Nursing Students' Knowledge Level Regarding Safe Medication Practices

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, Dr., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data may be requested from authors, but will not be shared in a database or on any site.